CLINICAL TRIAL: NCT03884543
Title: Driving Pressure During General Anesthesia for Open Abdominal Surgery (DESIGNATION) - a Randomized Clinical Trial
Brief Title: Driving Pressure During General Anesthesia for Open Abdominal Surgery
Acronym: DESIGNATION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Amsterdam UMC, location VUmc (Other); Noord West Ziekenhuizen location Alkmaar (Unknown); University Medical Center Groningen (Other); Radboud University Medical Center (Other); HagaZiekenhuis (Other); Rijnstate Hospital (Other); Medical Center Haaglanden (Other); Bernhoven Hospital (Other); Onze Lieve Vrouwe Gasthuis (Other); Albert Schweitzer Hospital (Other); Frisius Medisch Centrum (Other); Leiden University Medical Center (Other); Maastricht University Medical Center (Other); Martini Hospital Groningen (Other); Erasmus Medical Center (Other); Spaarne Gasthuis (Other); University Hospital Carl Gustav Carus (Other); Bermanntrost BG Klinikum Halle (Unknown); Heinrich-Heine University, Duesseldorf (Other); Ospedale Policlinico San Martino (Other); Jeroen Bosch Ziekenhuis (Other); Meander Medical Center (Other); Isala (Other); Alrijne Hospital (Other); Antoni van Leeuwenhoek Ziekenhuis (Unknown); Medisch Spectrum Twente (Other); Campus Bio-Medico University (Other); Istituto Nazionale Tumori IRCCS - Fondazione G. Pascale (Network); University of Roma La Sapienza (Other); University of Campania Luigi Vanvitelli (Other); Hospital Universitario La Fe (Other); Medical University Innsbruck (Other)
Responsible Party: Principal Investigator, Prof. Dr. Marcus J. Schultz, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DESIGNATION
Record Dates: First submitted 2018-11-02; First posted 2019-03-21 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Postoperative Respiratory Complication
Keywords: Mechanical ventilation; Positive end-expiratory pressure; Driving pressure; Post-operative postoperative complications; Open abdominal surgery; Recruitment maneuver; PEEP

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individualized high PEEP strategy (Experimental): Recruitment maneuver (performed after induction of anesthesia, after any disconnection from the mechanical ventilator, and before extubation) followed by the decremental PEEP trial to determine the highest level of PEEP resulting in the lowest driving pressure. This is again followed by a recruitment maneuver, after which PEEP is set at the level indicated by the decremental PEEP trial.
  Interventions: Procedure: Individualized high PEEP strategy
- Standard low PEEP strategy (No Intervention): PEEP at maximum 5cm H2O. No recruitment maneuvers. Patients are randomized and intraoperatively ventilated with conventional strategy. (PEEP at maximum 5cm H2O without recruitment maneuvers)

INTERVENTIONS:
Procedure: Individualized high PEEP strategy — Patients are randomized and intra-operatively ventilated with an individualized high PEEP strategy (Highest PEEP with the lowest driving pressure with recruitment maneuvers)
  Arms: Individualized high PEEP strategy

SUMMARY:
The purpose of this international multicenter, patient and outcome-assessor blinded randomized controlled trial is to determine whether the application of an individualized high PEEP strategy, aiming at avoiding an increase in the driving pressure during intraoperative ventilation, protects against the development of postoperative pulmonary complications.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for open abdominal surgery
* High or intermediate risk for postoperative pulmonary complications according to ARISCAT score [J.Canet et al, Anesthesiology 2010;113]
* General anesthesia

Exclusion Criteria:

* Laparoscopic surgery
* Surgery in prone or lateral position
* Combined procedure with open abdominal and intrathoracic surgery
* Body mass index > 40 kg/m2;
* Reported pregnancy;
* Mechanical ventilation > than 30 minutes (e.g., in cases of general anesthesia because of surgery) within last 30 days;
* Any major previous lung surgery;
* History of previous severe chronic obstructive pulmonary disease (COPD) GOLD III or IV, or with (noninvasive) ventilation and/or oxygen therapy at home;
* (previous) acute respiratory distress syndrome (ARDS);
* Expected to require postoperative mechanical ventilation;
* Persistent hemodynamic instability or intractable shock;
* Severe cardiac disease (New York Heart Association class III or IV, or acute coronary syndrome, or persistent ventricular tachyarrhythmia's);
* Consented for another interventional study during anesthesia or refusal to participate in the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1468 (Actual)
Dates: Start 2019-04-23 (Actual); Primary Completion 2025-03-11 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Proportion of participants developing one or more postoperative pulmonary complications (PPCs) | The first 5 postoperative days
  Severe respiratory failure; ARDS; Suspected pulmonary infection; Pulmonary infiltrate ; Pleural effusion; Atelectasis; Pneumothorax; Bronchospasm; Aspiration pneumonitis; Cardiopulmonary edema

SECONDARY OUTCOMES:
Rate of mild respiratory failures | The first 5 postoperative days
  Defined as a PaO2 < 60 mmHg (or < 7.9 kPa) or SpO2 < 90% in room air, but responding to supplemental oxygen (excluding hypoventilation)
Proportion of participants developing one or more post-operative extra-pulmonary complications | The first 5 postoperative days
  Including sepsis (according to the SEPSIS-3 definition), septic shock (defined as sepsis with persisting hypotension requiring vasopressors to maintain MAP ≥ 65mmHg and having a serum lactate level >2 mmol/L despite adequate volume resuscitation), extra-pulmonary infection (including wound infection and any other infection), anastomic leak and acute renal failure (as defined by AKIN [Mehta RL., et al., Acute Kidney Injury Network: report of an initiative to improve outcomes in acute kidney injury. Crit Care, 2007])
Rate of intra-operative complications | For the length of the anesthesia, which will be estimated 2 to 5 hours.
The total amount and type of intraoperative fluid administration | For the length of the anesthesia, which will be estimated 2 to 5 hours
  Type of fluids: colloids, crystalloids or blood products
Rate of all-cause mortality and in-hospital mortality | Postoperative day 5, day 30 and day 90
Length of hospital stay | From the day of surgery until the day of discharge, up to day 90
Number of participants with an unscheduled Intensive Care Unit (ICU) (re-) admission and length of stay in Intensive care unit | From the day of surgery until the day of discharged, up to day 90
Assessment of postoperative wound healing | The first 5 postoperative days
  Visual inspection of the following: impairment of wound healing and/or wound infection;

CONTACTS AND LOCATIONS:
Overall Officials: Marcus J. Schultz, MD PhD, Principal Investigator — Department of Intensive Care; Markus W. Hollmann, MD PhD, Principal Investigator — Department of Anesthesiology
Locations (22):
- Germany (3):
  - University hospital Carl Gustav Carus, Dresden
  - Heinrich-Heine University Hospital Dusseldorf, Düsseldorf
  - Bermanntrost BG Klinikum Halle, Halle
- Italy (2):
  - Ospedale Policlinico San Martino, Genoa
  - University hospital Napoli, Napoli
- Netherlands (17):
  - Noordwest ziekenhuizengroep Alkmaar, Alkmaar
  - Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA), Amsterdam
  - Amsterdam UMC location VUmc, Amsterdam
  - Onze Lieve Vrouwen Gasthuis, Amsterdam
  - Rijnstate Hospital, Arnhem
  - Albert Schweitzer Ziekenhuis, Dordrecht
  - Martini Hospital, Groningen
  - UMC Groningen, Groningen
  - Spaarne Gasthuis Hospital, Haarlem
  - Medical Center Leeuwarden, Leeuwarden
  - Leiden UMC, Leiden
  - Maastricht UMC, Maastricht
  - Radboud UMC, Nijmegen
  - Erasmus Medisch Centrum, Rotterdam
  - Haaglanden Medisch Centrum, The Hague
  - HAGA, The Hague
  - Bernhoven Hospital, Uden

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Mehta RL, Kellum JA, Shah SV, Molitoris BA, Ronco C, Warnock DG, Levin A; Acute Kidney Injury Network. Acute Kidney Injury Network: report of an initiative to improve outcomes in acute kidney injury. Crit Care. 2007;11(2):R31. doi: 10.1186/cc5713. PMID 17331245
- [Derived] Writing and Steering Committees for the DESIGNATION-Investigators; Dorland G, Gama de Abreu M, Hemmes SNT, Hol L, Hollmann MW, van Meenen DMP, Nijbroek SGLH, Schultz MJ, Serpa Neto A, Vermeulen TD. Intraoperative Driving Pressure-Guided High PEEP vs Standard Low PEEP for Postoperative Pulmonary Complications. JAMA. 2025 Dec 3:e2523373. doi: 10.1001/jama.2025.23373. Online ahead of print. PMID 41334859
- [Derived] DESIGNATION-investigators. Driving Pressure During General Anesthesia for Open Abdominal Surgery (DESIGNATION): study protocol of a randomized clinical trial. Trials. 2020 Feb 18;21(1):198. doi: 10.1186/s13063-020-4075-z. PMID 32070400

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-01-12): https://cdn.clinicaltrials.gov/large-docs/43/NCT03884543/SAP_001.pdf